CLINICAL TRIAL: NCT03412721
Title: A Split-mouth Clinical Study on the Effectiveness of Er:YAG Pulse Therapy for Achieving Pre-emptive Dental Analgesia in Children
Brief Title: Effectiveness of Er:YAG Pulse Therapy for Achieving Pre-emptive Dental Analgesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PlovdivMU
Record Dates: First submitted 2018-01-08; First posted 2018-01-26 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2018-08

CONDITIONS: Caries, Dental
Keywords: laser analgesia; pediatric dentistry
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Split-mouth assignment with two-way repeated measures design Masking: Double (Participant, Outcomes Assessor)
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser analgesia (Experimental): Procedure: Laser analgesic procedure Performing protocol for pre-emptive laser analgesia with Er:YAG laser (Litetouch, Syneron) switched on.
  Interventions: Procedure: Laser analgesic procedure
- Placebo analgesia (Placebo Comparator): Procedure: Placebo analgesic procedure Performing imitation of laser analgesic protocol with Er:YAG laser (Litetouch, Syneron) switched off - no pulse energy applied.
  Interventions: Procedure: Placebo analgesic procedure

INTERVENTIONS:
Procedure: Laser analgesic procedure — Water mist spray set to "maximum", non-contact handpiece with sapphire tip. Tip-to-tissue distance 10 mm from the tooth neck, achieved by using a spacer. Energy is delivered to the enamel above the gingival margin adjacent to the cemento-enamel junction (perpendicularly towards the dental pulp) on each of the four line angles of the tooth for 30s, moving the laser handpiece in a sweeping action. Pulse energy - 0.2 W/ 10 Hz/ 20 mJ. Follows increase of energy and repetition of protocol - 0.6 W/ 15 Hz/ 40 mJ. Total duration of LA-induction - 240s.
  Arms: Laser analgesia
Procedure: Placebo analgesic procedure — Performing imitation of laser analgesic procedure. No pulse energy applied, non-contact handpiece with sapphire tip. Moving the laser handpiece in a sweeping action towards the cemento-enamel junction (pointing perpendicularly towards the dental pulp) on each of the four line angles of the tooth. Total duration of placebo analgesia induction - 240s.
  Arms: Placebo analgesia

SUMMARY:
The aim of this study is to determine the effectiveness of Er:YAG pulse therapy for achieving pulpal analgesia in pediatric patients and to quantify the duration and extent of any effects assessed.

Design: a randomized split-mouth study with two-way repeated measures design.

DETAILED DESCRIPTION:
The intention of the technique of "pre-emptive laser analgesia" is to reduce sensation in that small percentage of patients who may experience unpleasant sensations during caries removal. Laser analgesia is a non-invasive, non-thermogenic bio-modulation of the dental pulp reactivity aiming for reduction of impulse formation of the pulpal nociceptors. It is based on the idea that parallel with the ablative high-energy level laser action, simultaneous low level laser therapy (LLLT) may occur. We hypothesize that when operating at pulse energies below the Er:YAG laser ablation threshold of tooth structure, the laser energy leads to loss of impulse conduction of type A-delta nerve fibers in the dental pulp, leading to an analgesic effect.

ELIGIBILITY:
Exclusion criteria:

* Children who are considered medically compromised or medically complex patients. The absence of disease is confirmed by anamnestic interview with a parent or a care-giver of the child and excludes general acute or chronic disease, cognitive impairment, psychogenic nonepileptic events, radiotherapy in the maxillofacial region due to malignant process.
* Patients who are undergoing therapy with neurological, sedative, analgesic and/or anti-inflammatory drugs 7 days prior to treatment.
* Children, who are first time ever dental patients.

Inclusion criteria:

* Patients, identified as positive or definitely positive through Frankl behavioral rating scale.
* Patients who are not undergoing treatment or have been treated 6 months prior to inclusion with remineralizing agents.
* Patients, requiring conservative treatment of occlusal, caries on foramen caecum, and/or proximal caries on two first permanent upper jaw molars without prior restorations or dental sealants. Lesions are to be classified as moderate caries by the International caries detection and assessment system (ICDAS) with code 03 or code 04, which do not present spontaneous unprovoked pain, percussion or palpation pain or other symptoms, indicating of pulpal pathology. Included are carious lesions only on vital teeth, involving up to half of the dentine thickness, with no periodontal pathology. Laser fluorescence diagnosis of adjacent lesions with DIAGNODENT is limited to 20 - 35 scores included.
* Included are first molars which are not affected by hypoplasia or hypomineralization.

Obtained informed consent from parents or gave-givers to participate in the study, in which laser treatment and study procedures are explained in appropriate manner.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-09-08 (Actual)

PRIMARY OUTCOMES:
Pain felt during treatment according to a visual analogue scale | 1 hour
  Reported by the patient at the end of the dental treatment session on a VAS (visual analogue scale), which contains a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, which includes pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst'). The combination allows children to pick a facial expression, that corresponds with their pain and see a number that matches it.

SECONDARY OUTCOMES:
Changes in pulpal sensibility to electrical stimuli by electrical pulp tester | 25 minutes
  Evaluated via electrical pulp tester (EPT) 5 minutes before and on the 5th and 20th minute after laser/placebo analgesic procedure. EPT result is a number.
Changes in pulpal sensibility to cold-stimuli by a visual analogue scale | 25 minutes
  Cold-test is applied 4 minutes before and on the 6th and 21st minute after laser/placebo analgesia. Pain is reported by the patient on a VAS (visual analogue scale), which contains a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, which includes pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst').
Patient experience during analgesic or placebo procedure | 5 minutes
  evaluated by a patient questionnaire
Pain related behavior evaluated by the Faces, Legs, Activity, Cry, Consolability Behavioral Pain Rating Scale | 1 hour
  Evaluated by the outcomes assessor. The FLACC scale has five criteria - Faces, Legs, Activity, Cry, Consolability, which are each assigned a score of 0, 1 or 2. Total score of scale is summed in range 0 to 10, where: 0=relaxed and comfortable; 1-3=mild discomfort; 4-6=moderate pain; 7-10=severe pain.
Dynamics of the heart rate of the patient | 1 hour
  registered throughout the experiment via pulse oximeter
Need for local anesthesia infiltration during the treatment | 1 hour
  Registered with 1=no; 2=yes. Patients who request that the procedure is terminated to administer an anesthetic injection, are asked to rate their level of pain, according to aforementioned visual analogue scale, immediately following termination. The visual analogue scale contains a combination of Numeric Rating Scale (0-10, where 0 means no pain, 10 - worst possible pain) and Wong-Baker Faces Pain Scale, which includes pictures of facial expressions with correlating numbers of 0-10 (0 being 'no hurt' and 10 being 'hurts worst').

CONTACTS AND LOCATIONS:
Overall Officials: Elitsa Veneva, DMD, Principal Investigator — Medical University - Plovdiv, Bulgaria
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dental Medicine, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Veneva E, Raycheva R, Belcheva A. Efficacy of erbium-doped yttrium aluminium garnet for achieving pre-emptive dental laser analgesia in children: A study protocol for a randomized clinical trial. Medicine (Baltimore). 2018 Dec;97(51):e13601. doi: 10.1097/MD.0000000000013601. PMID 30572467